CLINICAL TRIAL: NCT04088409
Title: An Open-label, Active-Controlled, Safety, and Efficacy Study of Oral Baricitinib in Patients From 2 Years to Less Than 18 Years Old With Active Juvenile Idiopathic Arthritis-Associated Uveitis or Chronic Anterior Antinuclear Antibody-Positive Uveitis
Brief Title: A Study of Baricitinib (LY3009104) in Participants From 2 Years to Less Than 18 Years Old With Active JIA-Associated Uveitis or Chronic Anterior Antinuclear Antibody-Positive Uveitis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16277; I4V-MC-JAHW (Other: Eli Lilly and Company); 2019-000119-10 (EudraCT Number)
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis | interventions — baricitinib; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Baricitinib (Experimental): Participants ≥9 to <18 years of age were administered 4 milligrams (mg) baricitinib once daily (QD). Participants <9 years of age were administered 2 mg baricitinib QD.
  Participants <6 years of age received an oral suspension. Participants ≥6 to <12 years of age had the option of receiving an oral suspension. Participants >12 years of age were supplied tablets.
  Interventions: Drug: Baricitinib
- Adalimumab (Active Comparator): Participants received adalimumab administered subcutaneously (SC) once every 2 weeks. The dose was based on body weight: 20 mg every 2 weeks for participants weighing <30 kilograms (kg), or 40 mg every 2 weeks for participants weighing ≥30 kg.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104
  Arms: Baricitinib
Drug: Adalimumab — Administered SC
  Arms: Adalimumab

SUMMARY:
The reason for this study is to see if the study drug baricitinib given orally is safe and effective in participants with active juvenile idiopathic arthritis (JIA)-associated uveitis or chronic anterior antinuclear antibody-positive uveitis from 2 years to less than 18 years old.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of JIA-U or chronic anterior antinuclear antibody (ANA) positive uveitis without systemic features.
* Participants must have active anterior uveitis, defined as cellular infiltrate in the anterior chamber of SUN criteria grade ≥1+ at screening and randomization, despite prior treatment with adequate doses of topical steroid therapy and methotrexate (MTX).
* Participants must have an inadequate response or intolerance to MTX.
* Participants must be on a stable dose of corticosteroid eye drops for at least 2 weeks prior to screening with a maximum of 4 drops/day/eye at screening.
* Participants and their partners of child bearing potential must agree to use 2 effective methods of contraception for the duration of the study and for at least 1 week following the last dose of investigational product.

Exclusion Criteria:

* Participants must not have a history or presence of any autoimmune inflammatory condition other than JIA, such as Crohn's disease or ulcerative colitis.
* Participants must not have any contraindications to adalimumab.

  * Exception: Participants who are biologic disease-modifying antirheumatic drug (bDMARD) inadequate response or intolerance with a contraindication to adalimumab may be enrolled, as they will be assigned to baricitinib.
* Participants must not have increased intraocular pressure ≥25 millimeters of mercury (mm Hg) or that required treatment, including increases in medications, surgery, or hospitalization, within 4 weeks prior to baseline that, in the opinion of the investigator, would pose an unacceptable risk to the participant.
* Participants must not have had intraocular surgery within the 3 months prior to screening (such as for cataract(s), glaucoma or vitrectomy).
* Participants must not have a current or recent (<4 weeks prior to baseline) infection.
* Participants must not have a positive test for hepatitis B virus (HBV) at screening.
* Participants must not have evidence of active tuberculosis (TB) or untreated latent TB.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2028-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (20):
- France (3):
  - Hôpitaux Universitaires Paris Sud - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Universitaire Necker Enfants Malades, Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
- Germany (4):
  - Asklepios Klinik Sankt Augustin, Sankt Augustin, North Rhine-Westphalia
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Charité Campus Virchow-Klinikum, Berlin
  - Praxis Kinder- und Jugendrheumatologie Dr. Ivan Foeldvari, Hamburg
- Italy (2):
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Azienda Ospedaliero Universitaria Meyer, Florence
- Spain (4):
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona
  - Hospital Infantil Universitario Niño Jesús, Madrid, Madrid, Comunidad de
  - Hospital Universitario La Paz, Madrid, Madrid, Comunidad de
  - Hospital Universitario La Fe de Valencia, Valencia
- United Kingdom (7):
  - Bristol Royal Hospital for Children, Bristol, Bristol, City of
  - Cambridge Clinical Research Facility, Cambridge, Cambridgeshire
  - Alder Hey Children's Hospital, Liverpool, England
  - Royal Victoria Infirmary, Newcastle upon Tyne, England
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Great Ormond Street Hospital For Children NHS Foundation Trust, London
  - Sheffield Children's Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Ramanan AV, Guly CM, Keller SY, Schlichting DE, de Bono S, Liao R, Quartier P. Clinical effectiveness and safety of baricitinib for the treatment of juvenile idiopathic arthritis-associated uveitis or chronic anterior antinuclear antibody-positive uveitis: study protocol for an open-label, adalimumab active-controlled phase 3 clinical trial (JUVE-BRIGHT). Trials. 2021 Oct 9;22(1):689. doi: 10.1186/s13063-021-05651-5. PMID 34627340
- See also: A Study of Baricitinib (LY3009104) in Participants From 2 Years to Less Than 18 Years Old With Active JIA-Associated Uveitis or Chronic Anterior Antinuclear Antibody-Positive Uveitis — https://trials.lillytrialguide.com/en-US/trial/5MwLoOOn4GIPFAxy1iilv6

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 30 participants were enrolled in the study. One participant (in baricitinib arm) withdrew from the study before administration of the study drug. This study is conducted in 2 parts. Part A (24 weeks) and Part B (260 weeks). Participants assigned to baricitinib and completed the Part A as a responder continued receiving baricitinib until the end of study or discontinuation from the study.
Period: Part A
Arm/Group | Baricitinib | Adalimumab
Started | 25 | 5
Received At Least 1 Dose of Study Drug | 24 | 5
Completed | 10 | 0
Not Completed | 15 | 5
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Did Not Meet Randomization Criteria | 2 | 0
Not completed — Lack of Efficacy | 9 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Per Protocol, Participants in the Adalimumab Group Discontinued the Study | 0 | 4
Period: Part B
Arm/Group | Baricitinib | Adalimumab
Started | 10 | 0
Completed | 0 | 0
Not Completed | 10 | 0
Not completed — Ongoing Treatment | 10 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Baricitinib: Participants ≥9 to <18 years of age were administered 4 mg baricitinib QD. Participants <9 years of age were administered 2 mg baricitinib QD.
  Participants <6 years of age received an oral suspension. Participants ≥6 to <12 years of age had the option of receiving an oral suspension. Participants >12 years of age were supplied tablets.
- Adalimumab: Participants received adalimumab administered SC once every 2 weeks. The dose was based on body weight: 20 mg every 2 weeks for participants weighing <30 kg, or 40 mg every 2 weeks for participants weighing ≥30 kg.
- Total: Total of all reporting groups
Arm/Group | Baricitinib | Adalimumab | Total
Number analyzed (Participants) | 24 | 5 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.60 (3.53) | 6.60 (2.51) | 10.70 (3.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 5 | 19
  Male | 10 | 0 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 12 | 4 | 16
  Unknown or Not Reported | 10 | 1 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 20 | 4 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  France | 4 | 0 | 4
  Germany | 1 | 1 | 2
  Italy | 3 | 2 | 5
  Spain | 3 | 0 | 3
  United Kingdom | 13 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: Part A: Percentage of Responders for Baricitinib at Week 24
Description: Response was defined according to the Standardization of Uveitis Nomenclature (SUN) criteria as a 2-step decrease in the level of inflammation (anterior chamber cells) or decrease to zero through week 24, in the eye most severely affected at baseline.
Time Frame: Week 24
Population: All participants who received at least one dose of baricitinib in Part A.
Measure: Number; unit: Percentage of participants
Arm/Group | Baricitinib
Number analyzed (Participants) | 24
Percentage of participants | 33.3

2. Secondary Outcome: Change From Baseline in SUN Grade of Cells in the Anterior Chamber in the Most Severely Affected Eye
Description: Change from Baseline in SUN Grade of Cells in the Anterior Chamber in the Most Severely Affected Eye. Outcome data will be provided after the study is completed.
Time Frame: Baseline, Week 24
Reporting Status: Not Posted, anticipated posting 2029-07

3. Secondary Outcome: Change From Baseline in SUN Grade of Cells in the Anterior Chamber in the Less Severely Affected Eye (If Applicable)
Description: Change from Baseline in SUN Grade of Cells in the Anterior Chamber in the Less Severely Affected Eye (If Applicable). Outcome data will be provided after the study is completed.
Time Frame: Baseline, Week 24
Reporting Status: Not Posted, anticipated posting 2029-07

4. Secondary Outcome: Percentage of Responders in Participants With Bilateral Uveitis Disease at Baseline
Description: Response is defined according to the SUN criteria as a 2-step decrease in the level of anterior chamber cells in the most severely affected eye at baseline (or both eyes if the inflammation grade is the same in both eyes) and a 1-step decrease in the level of anterior chamber cells in the less severely affected eye at baseline. Outcome data will be provided after the study is completed.
Time Frame: Week 24
Reporting Status: Not Posted, anticipated posting 2029-07

5. Secondary Outcome: Change From Baseline in Visual Acuity Measured by Age-Appropriate Logarithm of the Minimum Angle of Resolution (LogMAR) Test
Description: Change from Baseline in Visual Acuity Measured by Age-Appropriate LogMAR Test. Outcome data will be provided after the study is completed.
Time Frame: Baseline, Week 24
Reporting Status: Not Posted, anticipated posting 2029-07

6. Secondary Outcome: Change From Baseline in Vitreous Haze
Description: Change from Baseline in Vitreous Haze. Outcome data will be provided after the study is completed.
Time Frame: Baseline, Week 24
Reporting Status: Not Posted, anticipated posting 2029-07

7. Secondary Outcome: Change From Baseline in Grade of Flare in the Anterior Chamber
Description: Change from Baseline in Grade of Flare in the Anterior Chamber. Outcome data will be provided after the study is completed.
Time Frame: Baseline, Week 24
Reporting Status: Not Posted, anticipated posting 2029-07

8. Secondary Outcome: Percentage of Participants With Inactive Anterior Uveitis (Using SUN Definition)
Description: Percentage of Participants with Inactive Anterior Uveitis (using SUN Definition). Outcome data will be provided after the study is completed.
Time Frame: Week 24
Reporting Status: Not Posted, anticipated posting 2029-07

9. Secondary Outcome: Time to Inactive Anterior Uveitis Disease (Using SUN Definition)
Description: Time to Inactive Anterior Uveitis Disease (Using SUN Definition). Outcome data will be provided after the study is completed.
Time Frame: Baseline through Week 24
Reporting Status: Not Posted, anticipated posting 2029-07

10. Secondary Outcome: Percentage of Participants Who Are Able to Taper Concomitant Topical Corticosteroids to <2 Drops Per Day
Description: Percentage of Participants who are Able to Taper Concomitant Topical Corticosteroids to <2 Drops Per Day. Outcome data will be provided after the study is completed.
Time Frame: Week 24
Reporting Status: Not Posted, anticipated posting 2029-07

11. Secondary Outcome: Pediatric American College of Rheumatology (PediACR30) Response Rate (For Participants With JIA-U)
Description: PediACR30 Response Rate (For Participants with JIA-U). Outcome data will be provided after the study is completed.
Time Frame: Week 24
Reporting Status: Not Posted, anticipated posting 2029-07

12. Secondary Outcome: Change From Baseline in Overall Uveitis-Related Disability
Description: Change from Baseline in Overall Uveitis-Related Disability. Outcome data will be provided after the study is completed.
Time Frame: Baseline, Week 24
Reporting Status: Not Posted, anticipated posting 2029-07

ADVERSE EVENTS:
Time Frame: Baseline Up To 55 Weeks
Description: All participants who received at least one dose of study drug.
Arm/Group | Baricitinib | Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/24 | 1/5
Other Adverse Events (participants affected / at risk) | 16/24 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baricitinib (N=24) | Adalimumab (N=5)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baricitinib (N=24) | Adalimumab (N=5)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Illness (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Bilirubin conjugated increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1) | 1 (1)
Mean platelet volume decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Bone development abnormal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-06-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT04088409/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-13): https://cdn.clinicaltrials.gov/large-docs/09/NCT04088409/SAP_001.pdf